CLINICAL TRIAL: NCT05860218
Title: A Suggested Functional Exercises Program For Patients With Chronic Mechanical Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Doha Ali Amin Ahmed (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, Doha Ali Amin Ahmed, principal investigator, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: mechanical low back pain
Record Dates: First submitted 2023-04-24; First posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Chronic Mechanical Low Back Pain
MeSH Terms: interventions — Counseling; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- advices (Other): • Group I (control) will receive advices only.
  Interventions: Other: advices
- exercises plus advices (Experimental): • Group II (experimental) will receive a suggested functional exercise program plus advises
  Interventions: Other: advices; Other: exercises plus advices

INTERVENTIONS:
Other: advices — The following advice will be given to the patients :
  1. Walking as flexibly (normally) as possible
  2. Advise when lifting ;
     * avoid twisting and bending.
     * for heavy objects use thighs with a vertical back.
     * at other times, use the back and flex it.
  3. Heat application for 20 mins twice /day .
  4. Avoid sitting or standing for prolonged period and change position every 15 mins.
  5. Sitting: Sit with a back support
  6. Driving: Use a back support (lumbar roll) at the curve of your back.
  7. Sleeping and lying down: Select a firm mattress and box spring set that does not sag. If necessary, place a board under your mattress. You can also place the mattress on the floor temporarily if necessary.
Other: exercises plus advices — In addition to the same advice of group A, a suggested functional exercise will be performed for this group.
  1. Sidestepping against band resistance:
  2. The quadriped opposite arm leg aganist resistance .
  3. Squat row on a balance board with band resistance:
  4. Front raise single leg support with band resistance:
  5. The Advanced Prone Bridge:
  6. Side sliding on a fitter board (lateral lunge with band):
  Other Names: a suggested functional exercise program plus advises.
  Arms: exercises plus advices

SUMMARY:
The aim of this study will be to investigate the effect of functional exercise on pain, functional disability and core strength in patients with chronic mechanical low back pain .

DETAILED DESCRIPTION:
To our knowledge, there has been not enough studies that investigated the effect of core strengthening by functional exercise on pain, functional disability and core muscle strength in patients with chronic mechanical low back pain. Therefore, this study may open up ways to other researchers to investigate and build up on this effect if present and address such an important issue.

the finding of this proposed work may help patients with chronic mechanical low back pain by addressing their pain, functional limitation, and/or participation restrictions. Consequently, this can speed up their recovery, return to work, decrease cost of treatment, improve psychological status, decrease level of irritability, and improve overall quality of life.

Patients with chronic mechanical low back pain will be recruited after approval of ethical committee of the faculty of physical therapy, Cairo University. All participants will sign a written informed consent form.

The subjects will be randomly assigned into one of two groups:

* Group I (control) will receive advices only.
* Group II (experimental) will receive a suggested functional exercise program plus advises.

the measurments will take before and after treatment programe .

ELIGIBILITY:
Inclusion Criteria:

* Chronic mechanical low back pain and their age will be ranged from 20 -45 years.
* History of chronic low back pain (≥3 months).
* Patients with Body Mass Index (BMI) between 18-28

Exclusion Criteria:

* Age younger than 20 or older than 45 years of age.
* History of any surgical procedure in the back or the lower extremities
* Back pain secondary to known specific pathology (e.g. infection, tumor, osteoporosis, fracture, structural deformity, inflammatory disorder (e.g. ankylosing spondylitis) or cauda equine syndrome).
* Patient with lumbar instability including spondylolisthesis.
* Red flags (e.g. fever, unexplained weight loss, progressive weakness, radiation to lower limb, bowel and bladder dysfunction).
* Pregnancy.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
pain in lower back | change from max pain point in 1 month
  will be measured by The Numeric Pain Rating Scale (NPRS). it consists of The 11-point numeric scale ranges from '0' representing one pain extreme (e.g., "no pain") to '10' representing the other pain extreme (e.g., "pain as bad as you can imagine" or "worst pain imaginable .patients are asked to indicate the point along the line that best reflect their pain intensity .
functional disability | change in 1 month
  will be measured by Arabic version of Oswestry Disability Index (ODI) is a self-reported questionnaire consisting of 10 questions related to back function . Each question is answered on a 6-item Likert scale and is scored from 0 (minimum degree of difficulty in that activity) to 5 (maximum degree of difficulty). These questions assess the activities of daily living in patients with LBP. The questions in the index include pain intensity, personal care, lifting, walking, sitting, standing, sleeping, sex life, social life and travelling.
  The validity of Arabic version of ODI is good intra-observer reliability was excellent . The correlations of the ODI with the VAS pain scale, the Roland-Morris Low Back Pain Disability and the Quebec Back Pain Disability.
core muscles stability | change in 1 month
  The researcher will conduct a series of core stability tests before and after the core training program. Core stability tests has been reported to be highly reliable (ICC ≥ 0.98) and showed moderate to high correlation with one another (correation coefficient ranged from 0.4 to 0.8) , The following core tests will be used: trunk flexion test (McGill's test) , Trunk extension (Sorenson Test) , Side plank test and prone plank test .
lower limb function | change in 1 month
  will measured by Functional assessment using one legged hops test The most commonly used functional tests are a series of one-legged hops described by Noyes et al. (1991). The sensitivity of the single (49%), triple (50%), crossover (58%), and timed (52%) hop tests were reported by Noyes et al. (1991). The specificity was 97% and 94% for the timed and single hops, respectively

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
undecided